CLINICAL TRIAL: NCT04528056
Title: Pilot Study of the Safety and Efficacy of Sulfasalazine in Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: treatment of PAH
Record Dates: First submitted 2020-08-14; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sulfasalazine; ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ambrisentan+Sulfasalazine (Experimental)
  Interventions: Drug: Sulfasalazine; Drug: Ambrisentan
- Ambrisentan+Sulfasalazine's placebo (Active Comparator)
  Interventions: Drug: Ambrisentan; Drug: Sulfasalazine's placebo
- Ambrisentan's placebo+Sulfasalazine (Experimental)
  Interventions: Drug: Sulfasalazine; Drug: Ambrisentan's placebo
- Ambrisentan's placebo+Sulfasalazine's placebo (Placebo Comparator)
  Interventions: Drug: Sulfasalazine's placebo; Drug: Ambrisentan's placebo

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine is an anti-inflammatory and immunosuppressive drug
  Arms: Ambrisentan's placebo+Sulfasalazine; Ambrisentan+Sulfasalazine
Drug: Ambrisentan — Ambrisentan is one of the specific drug therapy for pulmonary arterial hypertension
  Arms: Ambrisentan+Sulfasalazine; Ambrisentan+Sulfasalazine's placebo
Drug: Sulfasalazine's placebo — Sulfasalazine's placebo is similar to Sulfasalazine in form and dosage
  Arms: Ambrisentan's placebo+Sulfasalazine's placebo; Ambrisentan+Sulfasalazine's placebo
Drug: Ambrisentan's placebo — Ambrisentan's placebo is similar to Ambrisentan in form and dosage
  Arms: Ambrisentan's placebo+Sulfasalazine; Ambrisentan's placebo+Sulfasalazine's placebo

SUMMARY:
Under placebo control, the investigators intend to evaluate the effectiveness and safety of anti-inflammatory therapy and/or targeted drug therapy for early treatment of patients with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is characterized by decompensated increase of pulmonary artery pressure owing to continuous progression of pulmonary vascular resistance and can ultimately cause right heart failure even death. At present, the treatment of pulmonary arterial hypertension is mainly the application of specific drug therapy. Specific drug therapy involves the three major pathways of endothelin, nitric oxide and prostacyclin. The main mechanisms of vasodilation and anti-proliferation are used to treat pulmonary arterial hypertension. However, the price of specific drug therapy is too expensive, which puts huge financial pressure on patients. Evidence shows that inflammation exists in the early stages of pulmonary arterial hypertension and anti-inflammatory treatment is effective in animal experiments. Under placebo control, the investigators intend to evaluate the effectiveness and safety of anti-inflammatory therapy and/or targeted drug therapy for early treatment of patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary artery systolic pressure estimated in the most recent echocardiography examination before screening ≧40mmHg.
2. Before the study, subjects received the best traditional pulmonary arterial hypertension(PAH) treatment (such as oral Ca2+ antagonists, oxygen therapy, digoxin, diuretics, and anticoagulants), and no increase, discontinuation, or dose change at least one month before randomization. But it is allowed to stop or adjust anticoagulants, and adjust the therapeutic dose of diuretics.
3. The results of echocardiography showed that the systolic and diastolic functions of the left ventricle were normal, and there was no clinically significant left heart disease (such as mitral valve disease).

Exclusion Criteria:

1. Patients who have received endothelin receptor antagonists and anti-inflammatory drugs within 30 days before randomization.
2. Patients with changes in the basic PAH treatment within one month before randomization (such as addition/removal of therapeutic drugs or dose adjustment; including but not limited to oxygen, diuretics, digoxin, anticoagulants, immunosuppressants, or Ca2+ antagonists ). But we allows the discontinuation of anticoagulants or change the dose and the change of diuretic dose.
3. Patients who diagnosed with other etiology of PAH, such as portal hypertension, pulmonary vein occlusive disease, etc.
4. Patients who have a history of left heart disease including ischemic heart disease, myocardial infarction, symptomatic coronary artery disease; or trans-channel radionuclide angiography, angiography, or echocardiography as assessed by mean pulmonary capillary wedge pressure (or left ventricular end diastolic volume) ≥ 15 mmHg or left ventricular ejection fraction ≤ 40%; or systemic hypertension that cannot be effectively controlled, systolic blood pressure> 160 mmHg or diastolic blood pressure> 100 mmHg.
5. Patients who have a history of lung diseases, including chronic obstructive pulmonary disease, interstitial lung disease, etc.
6. Patients who have a history of blood diseases, including a history of coagulation disorders within 6 months before screening.
7. Patients who are allergic to two or more drugs or food; or are known to be allergic to one anti-inflammatory drug (steroidal or non-steroidal anti-inflammatory drug).
8. Liver function test exceeds or equals 3 times the upper limit of normal or suffering from known Child-Pugh Class C liver disease.
9. Patients with chronic renal insufficiency, and the screening creatinine value is greater than 2.5mg/dL (221μmol/L) or need dialysis.
10. Patients with other diseases or conditions that can affect the results of the research.
11. Patients who participated in other study drugs or medical devices within 30 days before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Confirmed Clinical Adverse Event up to the End of Treatment | Up to end of treatment (data presented up to month 6)
  Clinical adverse event was defined as death.

SECONDARY OUTCOMES:
Change From Baseline to Month 6 in 6-minute Walk Distance | Baseline to month 6
  The 6-minute walk test (6MWT) is a non-encouraged test, performed in a 30 m long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. These guidelines were provided to all sites. For patients who had never performed a 6MWT previously, a training test was required before the qualifying tests for inclusion were performed.
Change From Baseline to Month 6 in Inflammation Factor | Baseline to month 6
  Compose of Interleukin-6
Change From Baseline to Month 6 in Echocardiography Examination | Baseline to month 6
  Assessment of pulmonary artery systolic pressure by echocardiography
Change From Baseline to Month 6 in Cardiac Function | Baseline to month 6
  Compose of B-type natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Jieyan Shen, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, China